IRB NUMBER: 02-18-58. IRB APPROVAL DATE: 2/4/2019 IRB EFFECTIVE DATE: 2/5/2019 IRB EXPIRATION DATE: 2/3/2020

# UNIVERSITY HOSPITALS CLEVELAND MEDICAL CENTER CONSENT FOR INVESTIGATIONAL STUDIES

**Project Title:** The Use of 3D Printed Models in Mohs Micrographic Surgery

Principal Investigator: Site PI:Dr. Margaret Mann MD; Research PI: Dr. Daniel Popkin MD, PhD

## Introduction/Purpose

Patients undergoing Mohs micrographic surgery frequently experience anxiety. It has been suggested that enhanced patient education prior to the procedure may decrease patient anxiety. The purpose of our study is to investigate if optimized patient education enhances patient understanding, decreases patient anxiety and increases patient satisfaction. If you would like to participate you will be asked to fill out several study questionnaires throughout your Mohs day, initially before surgery and following the first stage of your Mohs procedure. The pre-surveys & post-surveys will take only approximately 5 minutes each to complete. If you do not wish to participate please let us know.

## **Study Procedures**

Only 1 visit will be required to participate in this study. If you are eligible to participate, the following research procedures will be performed:

- 1. **Baseline Testing:** You will be asked to complete baseline surveys to assess your preoperative anxiety and understanding of Mohs surgery
- 2. Educational Intervention: You will be provided an explanation of Mohs surgery
- 3. **Post-Stage Testing:** Following the first stage of your Mohs surgery you will be asked to complete post-intervention surveys regarding your anxiety, understanding and satisfaction with the explanation of Mohs surgery provided to you

#### **Risks**

Questionnaires: There are no known risks associated with filling out questionnaires. However, some patients feel uncomfortable answering some of the questions. If you do not wish to answer a question, you may skip this question and move to the next one.

#### **Benefits**

There will be no direct benefit for your participation in this study. However, the information gained from this research may provide information about preoperative counselling that may help physicians the delivery of information regarding the Mohs procedure.

# **Alternatives to Study Participation**

The only alternative is to not participate. Your access to care and treatment will not be affected, should you decide you do not want to participate in this research study.

#### Compensation

There will be no compensation for your participation in this study.

### **Confidentiality**

We will not contact you again once the survey is completed. Please note that your name or any personal health information will not be connected to the survey and your surveys will be assigned an ID number. Answering this survey will not affect your health care at University Hospitals. You Version date 1.2.2019

Page 1 of 2

IRB NUMBER: 02-18-58.
IRB APPROVAL DATE: 2/4/2019
IRB EFFECTIVE DATE: 2/5/2019
IRB EXPIRATION DATE: 2/3/2020

# UNIVERSITY HOSPITALS CLEVELAND MEDICAL CENTER CONSENT FOR INVESTIGATIONAL STUDIES

**Project Title:** The Use of 3D Printed Models in Mohs Micrographic Surgery

Principal Investigator: Site PI:Dr. Margaret Mann MD; Research PI: Dr. Daniel Popkin MD, PhD

will not directly benefit from this study, however, we hope to this project will help us to better educate future Mohs patients. Your participation in this survey is voluntary and you can stop your participation at any time.

### **Contact information**

Mark Biro has described to you what is going to be done, the risks, hazards, and benefits involved. The Principal Investigator Dr. Mann can also be contacted at <a href="margaret.mann@uhhospitals.org">margaret.mann@uhhospitals.org</a>. If you have any questions, concerns or complaints about the study in the future, you may also contact them later.

Completion of the questionnaires indicates your consent for participation in this study

Version date 1.2.2019